CLINICAL TRIAL: NCT06265974
Title: ECHOQUALITY: Evaluation of Image Quality in Obstetrical Ultrasonography: Comparison Between Subjective Assessment and Contrast-to-noise Ratio
Brief Title: Evaluation of Image Quality in Obstetrical Ultrasonography: Comparison Between Subjective Assessment and Contrast-to-noise Ratio
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECHOQUALITY
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ultrasonography; Obstetrics
Keywords: Quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine whether the subjective assessment of the quality of obstetrical ultrasonography pictures can be similar to that of an objective tool.

The main question it aims to answer is:

Is the subjective assessment of the quality of obstetrical ultrasonography pictures by a young practitioner and an experienced one can be similar to that of an objective tool, such as the contrast-to-noise ratio (CNR)? The contrast-to-noise ratio is commonly used in radiology to evaluate image quality by assessing the ability to distinguish differences between two elements.

The investigators selected a retrospective cohort of 198 patients, including three pictures per fetus screened between 18 and 18 weeks and 6 days. For each picture, the investigators assessed the quality of two different elements and the entire image, and then calculated the CNR using software. The investigators will compare the three assessment between them

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent ultrasound between 18 weeks and 18 weeks + 6 days for prenatal diagnosis
* Ultrasound performed by the same practitioner
* Ultrasound performed on the same ultrasound machine "Voluson E10", with the "RM6C" probe

Exclusion Criteria:

* Patient's refusal
* Use of another ultrasound device other than the "Voluson E10", and/or an ultrasound probe other than the "RM6C"
* Intrauterine fetal deaths

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women having undergone an ultrasound between 18 weeks and 18 weeks + 6 days at the Multidisciplinary Prenatal Diagnostic Center of Poitiers University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
The comparability between a subjective and objective assessment of the contrast to noise ratio of an obstetric ultrasound image | baseline
  Both an experienced operator (a Ph.D. doctor) and a novice operator (a residency student) subjectively evaluated the contrast and noise of each region of interest previously chosen. Contrast was scored on a scale of 1 to 3, with 1 indicating low contrast, 2 for medium, and 3 for high contrast. Noise was scored on the same scale, with 1 corresponding to low noise, 2 for medium, and 3 for high noise. The subjective contrast to noise ratio (CNR) was determined by the ratio between these two scores.
  To assess the objective CNR, computer-assisted image analysis was performed using MATLAB software.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital La MILETRIE, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided